CLINICAL TRIAL: NCT05577780
Title: Femoral Neck Fracture Between 45 and 64 Years : Internal Fixation Versus Arthroplasty
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Mongi Slim Hospital (Other)
Responsible Party: Principal Investigator, mohamed hedi ezzine, Principal Investigator, medical doctor, assistant professor, Mongi Slim Hospital
Other Study IDs: mongislim1
Record Dates: First submitted 2022-09-27; First posted 2022-10-13 (Actual); Last update posted 2022-10-13 (Actual); Status verified 2022-10

CONDITIONS: Femoral Neck Fractures
MeSH Terms: conditions — Femoral Neck Fractures | interventions — Fracture Fixation, Internal; Arthroplasty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- internal fixation
  Interventions: Procedure: internal fixation
- arthroplasty
  Interventions: Procedure: internal fixation

INTERVENTIONS:
Procedure: internal fixation — Patients with femoral neck fractures are treated with pinning or hip arthroplasty, depending on the age of the patient and the presence and degree of displacement
  Other Names: arthroplasty

SUMMARY:
The therapeutic choice for femoral neck fracture is conventionally made between conservative treatment and total hip arthroplasty. This choice for patients aged between 45 and 64 years old remains a controversial subject.

The aim of our work was to describe the current situation in the management of femoral neck fractures in these patients and to evaluate the results of the two options

DETAILED DESCRIPTION:
Our study was retrospective descriptive including patients aged between 45 and 64 years operated between January 2015 and December 2022 for femoral neck fracture. The patients will be divided into two groups: The internal fixation group and the arthroplasty group . Epidemiological, clinical and radiological data as well as therapeutic results and postoperative complications will be analysed.

ELIGIBILITY:
Inclusion Criteria:

* Femoral neck fracture between 45 and 64 years

Ages: 45 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Femoral neck fracture between 45 and 64 years
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2015-01-10 (Actual); Primary Completion 2022-12-10 (Estimated); Study Completion 2023-01-10 (Estimated)

PRIMARY OUTCOMES:
The Parker Mobility Score | Baseline, Month 3
  The Parker Mobility Score answers three questions, each valued 0-3 points. Based on the sum of the mobility assessment in three different situations (able to get about the house, able to get out of the house and able to go shopping), the total score ranges from 0-9. For each of the three situations the mobility has to be scored on: no difficulty (3 points), with an aid (2 points), with help from another person (1 point) or not at all (0 points). The highest overall score of 9 indicates the best possible mobility
The Parker Mobility Score | Baseline, Month 6
  The Parker Mobility Score answers three questions, each valued 0-3 points. Based on the sum of the mobility assessment in three different situations (able to get about the house, able to get out of the house and able to go shopping), the total score ranges from 0-9. For each of the three situations the mobility has to be scored on: no difficulty (3 points), with an aid (2 points), with help from another person (1 point) or not at all (0 points). The highest overall score of 9 indicates the best possible mobility
GARDEN classification | Baseline
  Garden described particular femoral neck and acetabular trabeculae patterns which can assist in recognizing differences within this classification system
  Garden stage I: undisplaced incomplete, including valgus impacted fractures medial group of femoral neck trabeculae may demonstrate a greenstick fracture Garden stage II: undisplaced complete no disturbance of the medial trabeculae Garden stage III: complete fracture, incompletely displaced femoral head tilts into a varus position causing its medial trabeculae to be out of line with the pelvic trabeculae Garden stage IV: complete fracture, completely displaced femoral head aligned normally in the acetabulum and its medial trabeculae are in line with the pelvic trabeculae In general, stage I and II are stable fractures and can be treated with internal fixation (head-preservation) and stage III and IV are unstable fractures and hence treated with arthroplasty (either hemi- or total arthroplasty)
Postel Merle d'Aubigné score(PMA) | Baseline, Month 3
  the rating of Postel Merle D'Aubigné studies the pain, mobility and the walk and gives them a value from 0 to 6, allowing a global assessment of hip's function with a total of 18 marks for a normal hip. The PMA score is excellent if the score is 18, very good if the score is 17, good if the score is between 15 and 16, average if the score is between 13 and 14, poor if the score is between 9 and 12 and bad if the score is less than 9.
Postel Merle d'Aubigné score(PMA) | Baseline, Month 6
  the rating of Postel Merle D'Aubigné studies the pain, mobility and the walk and gives them a value from 0 to 6, allowing a global assessment of hip's function with a total of 18 marks for a normal hip. The PMA score is excellent if the score is 18, very good if the score is 17, good if the score is between 15 and 16, average if the score is between 13 and 14, poor if the score is between 9 and 12 and bad if the score is less than 9.